CLINICAL TRIAL: NCT04773782
Title: A Phase 1/2, Single-arm Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of Avapritinib in Pediatric Patients With Solid Tumors Dependent on KIT or PDGFRA Signaling
Brief Title: A Study of Avapritinib in Pediatric Patients With Solid Tumors Dependent on KIT or PDGFRA Signaling
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-3101
Record Dates: First submitted 2021-02-09; First posted 2021-02-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Unspecified, Child; Relapsed Solid Neoplasm; CNS Tumor
Keywords: KIT; PDGFRA; Relapsed/Refractory Solid Tumor; Glioma; H3K27M; DMG-H3K27a
MeSH Terms: conditions — Central Nervous System Neoplasms; Recurrence; Glioma | interventions — avapritinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- avapritinib (Experimental): Avapritinib tablets for oral administration. Avapritinib will be dosed daily for 28 day cycles.
  Interventions: Drug: avapritinib

INTERVENTIONS:
Drug: avapritinib — oral administration
  Other Names: BLU-285

SUMMARY:
This is a Phase 1/2, multicenter, open-label trial of avapritinib in participants 2 to < 18 years of age with advanced relapsed/refractory (R/R) solid tumors, including central nervous system (CNS) tumors, that harbor a PDGFRA and/or KIT mutation (including non-synonymous point mutations, insertions, and deletions) or amplification, or DMG-H3K27a who have no available curative treatment options. This is a single-arm trial in which all participants will receive avapritinib. The study consists of 2 parts: dose confirmation, safety, and PK (Part 1) and initial efficacy, safety, and PK at the Part 2 recommended dose (Part 2).

ELIGIBILITY:
Inclusion Criteria

1. Participant must be 2 to < 18 years of age at the time of signing the informed consent.
2. Diagnosis

   1. Participant has confirmed diagnosis of R/R solid tumor, including CNS tumors, with a mutation (including non-synonymous point mutations, insertions, and deletions) in PDGFRA and/or KIT (confirmed by local mutational testing of tumor sample) that has progressed despite standard therapy and no alternative treatment option is available. Participant with R/R solid tumors with only PDGFRA and/or KIT amplifications may be included with approval from the Sponsor.

      OR
   2. Participant has confirmed diagnosis of DMG-H3K27a (confirmed by local testing of tumor sample) that has failed standard therapy or for which no standard therapy that may convey clinical benefit exists, as judged by the investigator.
3. Participants with CNS disease should be on a stable (≤ 10% change) or decreasing dose of corticosteroids for at least 7 days prior to first dose of avapritinib, with no plans for dose escalation.
4. Disease extent: a. Part 1: All participants must have at least 1 measurable lesion as defined by RECIST v1.1 or Response Assessment in Neuro-Oncology (RANO) (for CNS tumors). If radiation therapy has been administered, at least 1 measurable lesion must not have been irradiated, or must have clearly progressed since being irradiated as per RANO and must be ≥ 12 weeks from radiation to any target lesion.

   b. Part 2: All participants must have at least 1 measurable lesion as defined by RECIST v1.1 or RANO (for CNS tumors). For Participants with DMG-H3K27a or PDGFRA and/or KIT mutant/amplified solid tumors, including CNS tumors that have progressed despite prior therapy, who have received radiation therapy, at least 1 measurable lesion must not have been irradiated, or must have clearly progressed since being irradiated as per RANO and must be ≥ 12 weeks from radiation to any target lesion. For up to 5 Participants with newly diagnosed DMG-H3K27a where there is no standard therapy that may convey clinical benefit exists as judged by the investigator, progression of disease of a measurable lesion after irradiation is not required.
5. A Lansky (< 16 years of age) or Karnofsky (≥ 16 years of age) score of at least 50. If the Participant is unable to walk due to paralysis, but is mobile in a wheelchair, the participant is considered ambulatory for the purpose of assessing their performance status.
6. Participant agrees to utilize contraception consistent with local regulations.

   * Male participants: Are vasectomized, or agree to use condoms, as defined in Section 5.4.2, from the start of Screening until 6 weeks after the last dose of study treatment, or practice true abstinence (when this is in line with the preferred and usual lifestyle of the Participant, see Section 5.4.2), or have a female partner who is NOT of childbearing potential.
   * Female participants: Agree to use effective contraception, as defined in Section 5.4.2, from the start of Screening until 6 weeks after the last dose of study treatment and have a male partner who uses a condom, or practice true abstinence (when this is in line with the preferred and usual lifestyle of the Participant), or have a male partner who is vasectomized with confirmed azoospermia.
7. Participant can give written informed consent/assent before any study-specific Screening procedures (if feasible). Parental/legal guardian consent will be determined by local, regional, and/or national guidelines.

Exclusion Criteria

1. Participant has any of the following within 14 days before the first dose of study treatment:

   1. Platelet count < 75 × 10^9/L (< 100 × 10^9/L if a CNS tumor) with no platelet transfusion within 14 days prior to the measurement.
   2. Absolute neutrophil count (ANC) < 1.0 × 10^9/L.
   3. Hemoglobin < 8.0 g/dL with no RBC transfusion ≤ 7 days prior to the measurement.
   4. AST or ALT > 3 × the ULN for age; except in Participants with tumor involvement of the liver who must not have AST and ALT > 5 × ULN for age.
   5. Total bilirubin > 1.5 × ULN for age; and in presence of Gilbert's syndrome, total bilirubin > 3 × ULN or direct bilirubin > 1.5 × ULN.
   6. Serum creatinine > 1.5 × ULN for age.
   7. International normalized ratio or prothrombin time (PT) > ULN (> 1.5 × ULN if on prophylactic reversible anticoagulants).
2. Participant has a QTcF > 470 msec. Participant has a familial or personal history of prolonged QT syndrome or Torsades de pointes.
3. Participant has clinically significant, uncontrolled cardiovascular disease including congestive heart failure Grade III or IV according to the New York Heart Association classification; myocardial infarction or unstable angina within the previous 6 months, uncontrolled hypertension (> 95th percentile for age), or clinically significant, uncontrolled arrhythmias, including bradyarrhythmias that may cause QT prolongation (eg, Type II second-degree heart block or third-degree heart block).
4. Participant received the following systemic antineoplastic therapies:

   1. Temozolomide within 4 weeks prior to the first dose of study drug
   2. Nitrosurea within 6 weeks prior to the first dose of study drug
   3. Any other systemic antineoplastic therapy (including experimental therapy) within 5 half-lives or 28 days prior to the first dose of study drug, whichever is shorter.
   4. Focal external beam radiotherapy, including stereotactic radiosurgery, within 6 weeks prior to the first dose of avapritinib to either target or nontarget lesions. Systemic radiopharmaceuticals, including nonstereotactic radiosurgery, within 2 weeks of the first dose of avapritinib (within 6 weeks for Participants with CNS tumors). Craniospinal irradiation within 6 weeks prior to the first dose of avapritinib.
   5. All AEs related to other antineoplastic therapies (eg, systemic antineoplastics, radiotherapy) must have resolved to Grade ≤ 1 (Grade ≤ 2 for peripheral neuropathy and/or ototoxicity) prior to the first dose of avapritinib.
5. Participant has previously received treatment with avapritinib.
6. Participant received autologous stem cell transplant following myeloablative therapy or chimeric antigen receptor T cell therapy within 3 months prior to the first dose of avapritinib or prior allogeneic stem cell transplant within 1 year and no evidence of Grade 1 or greater graft-versus-host disease and no immunosuppressants for graft-versus-host disease (steroids for primary malignancy being permitted). Participants who received stem cell reinfusion following nonmyeloablative therapy are eligible once they meet the peripheral blood count criteria in Exclusion Criterion #1.
7. Participant requires ongoing treatment or has received treatment within 28 days before the start of avapritinib administration with drugs or foods that are strong CYP3A inhibitors or inducers.
8. Participant has had a major surgical procedure within 14 days of the first dose of study treatment (procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures).
9. Participant has a history of another primary malignancy that has been diagnosed or required therapy within 3 years before the first dose of avapritinib. The following prior malignancies are not exclusionary: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site.
10. Female subjects of childbearing potential who are unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 6 weeks after the last dose of study treatment. Male subjects who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 6 weeks after the last dose of study treatment.
11. Participant is pregnant, as documented by a serum β-hCG pregnancy test consistent with pregnancy obtained at Screening and within 72 hours before the first dose of study treatment. Participants with β-hCG values that are within the range for pregnancy but are not pregnant (false-positives) may be enrolled with written consent of the Sponsor after pregnancy has been ruled out. Female subjects of nonchildbearing potential (premenarchal, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) do not require a serum β-hCG test.
12. Participant is breastfeeding.
13. Participant has prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the Participant; alter the absorption, distribution, metabolism, or excretion of the study drug; or impair the assessment of study results.
14. History of thrombosis requiring treatment within the past 6 months. This exclusion does not apply to catheter-related thrombosis if the catheter has been removed and did not require any other treatment in the previous 3 months.
15. Participants who require anticoagulants, with the exception of stable doses of prophylactic reversible anticoagulants.
16. Participants who are unable to swallow tablets (in Part 1) or minitablets (in Part 2) within the sprinkle capsules.
17. Participants with a known risk of intracranial bleeding, such as a brain aneurysm that has not been removed or repaired, or a history of intracranial bleeding within the past year, or radiographic evidence of hemorrhage on Screening MRI. Exceptions are: Participants with primary CNS tumors (provided they have not had CNS bleeding within 2 weeks of the first dose of avapritinib) or Participants with punctate hemorrhages < 3 mm.
18. History of a seizure disorder that is not well controlled on current antiepileptic medications.
19. Participant is unwilling or unable to comply with scheduled visits, treatment administration plan, laboratory tests, or other study procedures and study restrictions.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Determination of recommended Part 2 dose (Part 1) | up to 8 months
Objective Response Rate (Part 2) | up to 36 months
Rate and severity of adverse events (Part 1) | up to 8 months

SECONDARY OUTCOMES:
Objective Response Rate (Part 1 and Part 2) | up to 42 months
Rate and severity of adverse events (Part 1 and Part 2) | up to 42 months
Palatability assessments as measured by the 5-point Hedonic scale (Part 1 and Part 2) | up to 42 months
Duration of Response (Part 1 and Part 2) | up to 42 months
Progression-free survival (Part 1 and Part 2) | up to 42 months
Disease control rate (Part 1 and Part 2) | up to 42 months
Time to response (Part 1 and Part 2) | up to 42 months
Cmax (Part 1 and Part 2) | up to 36 months
AUC(0-24) (Part 1 and Part 2) | up to 36 months
Tmax (Part 1) | up to 36 months
T 1/2 (Part 1) | up to 36 months
Ctrough (Part 2) | up to 36 months
Change from baseline in levels of KIT and PDGFRA mutant allele fractions in peripheral blood (Part 1 and Part 2) | up to 42 months

CONTACTS AND LOCATIONS:
Locations (26):
- United States (15):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California San Francisco, Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Sydney Children's Hospital, Kids Cancer Center, Sydney, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
- Medizinische Universitat Wein, Vienna, Vienna, Austria
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Gustave Roussy, Villejuif, France
- Germany (2):
  - Universitaetsmedizin Göttingen, Göttingen, Lower Saxony
  - Hopp Children's Cancer Center, Heidelberg
- Dipartimento di Oncologia Medica ed Ematologia - S.C. Pediatria Oncologica, Milan, Italy
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medial Center, Seoul
- Great Ormond Street Hospital For Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No